CLINICAL TRIAL: NCT02183246
Title: A Phase III, Double-Blind, Randomized, Placebo-Controlled Study of Porfiromycin Used as an Adjuvant to Radiation Therapy in Postoperative Head and Neck Cancer Patients
Brief Title: Porfiromycin Used as an Adjuvant to Radiation Therapy in Postoperative Head and Neck Cancer Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1164.4
Record Dates: First submitted 2014-07-04; First posted 2014-07-08 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Head and Neck Neoplasms
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Porfiromycin; Radiotherapy

ARMS (2):
- Porfiromycin + Radiotherapy (Experimental)
  Interventions: Drug: Porfiromycin; Radiation: Radiotherapy
- Placebo + Radiotherapy (Placebo Comparator)
  Interventions: Drug: Placebo; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Porfiromycin
  Arms: Porfiromycin + Radiotherapy
Drug: Placebo
  Arms: Placebo + Radiotherapy
Radiation: Radiotherapy

SUMMARY:
Determination of efficacy and safety of porfiromycin versus placebo as an adjuvant to radiotherapy in postoperative head and neck a cancer patients as well as assessment of population pharmacokinetic parameters.

ELIGIBILITY:
Inclusion Criteria:

* Male or female postoperative radical neck surgery patients with histologically proven Stage III or IV (without distant metastases) epidermoid (squamous cell) carcinoma of the head and neck limited to the following locations as defined by the American Joint Commission (AJC): lip and oral cavity, pharynx, or larynx.
* Postoperative radical patients whose specimen had a) microscopic positive tumor cell margins (< 2mm from surgical margin) or b) extranodal capsular spread (perineural-vascular embolization) or c) two or more positive nodes
* Postoperative radical neck patients must have received Radiotherapy (RT).
* Performance status of ≥ 70 on the Karnofsky Performance Score (KPS) at screening.
* Patients ≥ 18 years of age
* Patients must have provided written informed consent prior to participation in the trial.
* Patients must have demonstrated an educational level and a degree of understanding such that they could communicate effectively with the investigator.

Exclusion Criteria:

* Patients that received any prior chemotherapy including mitomycin-C or porfiromycin.
* Treatment with granulocyte, granulocyte-macrophage stimulating factor (G-CSF, GM-CSF) or Interleukin-11 within 30 days prior to start of RT.
* RT within the treatment field for any malignancy within the past five years.
* Patients who had any gross (visible or palpable) residual disease left after surgery.
* Patients who met any of the following clinical laboratory criteria upon screening:

  1. Granulocyte (neutrophil) count of < 1,500/cubic millimeters (mm3)
  2. Platelets < 75,000/mm3
  3. Prothrombin time (PT) and partial thromboplastin time (PTT) > 1.5 times the upper limit of normal (ULN) in seconds.
* Women who were pregnant or nursing.
* Women of childbearing potential who were unwilling to utilise a medically acceptable method of contraception (oral contraceptives, intrauterine devices, diaphragm or subdermal implants eg: Norplant®).
* Other malignancies active within the past five years (other than basal or squamous cell carcinomas of the skin outside the planned radiation portals, or in situ carcinoma of the cervix).
* The presence of more than one primary tumor or presence of distant metastases.
* The presence of any other life-threatening illness, such a severe chronic lung, liver, or heart disease that would be expected to be fatal within five years, regardless of the patient's cancer status.
* Patients who participated in a clinical trial with another investigational drug or treatment 30 days prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2000-05; Primary Completion 2000-12 (Actual)

PRIMARY OUTCOMES:
Time to Disease Progression | week 4 and 8 post treatment, every 8 weeks until end of study
Maximum toxicity grades of Adverse Events (AE) | until 42 days after end of treatment
Time to non-accidental death | week 4 and 8 post treatment, every 8 weeks until end of study
Serum porfiromycin concentration-time profile | up to week 7

SECONDARY OUTCOMES:
Death for any reason | 4 weeks post treatment for every 8 weeks through 48 weeks, every 12 weeks until end of study
Loss of local or regional control, distant metastasis or death for any reason | 4 weeks post treatment for every 8 weeks through 48 weeks, every 12 weeks until end of study
Loss of local or regional control or distant metastasis | 4 weeks post treatment for every 8 weeks through 48 weeks, every 12 weeks until end of study
Loss of local or regional control | 4 weeks post treatment for every 8 weeks through 48 weeks, every 12 weeks until end of study
Occurrence of Adverse Events | up to week 16
Significant changes in laboratory tests | up to week 7
Changes from baseline in Patients health related Quality of life-Questionnaires | week 1, 5, 7, 4 weeks post treatment, every 12 weeks until end of study